CLINICAL TRIAL: NCT05465993
Title: An International Multi-institution Real-world Study of the Optimal Surveillance Frequency for Stage II/III Gastric Cancer
Brief Title: the Optimal Surveillance Frequency for Stage II/III Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director of gastric surgery, Fujian Medical University
Other Study IDs: GCFU-01
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; surveillance; cost-effectiveness; real-world study
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to lacking of evidence on surveillance for gastric cancer (GC), this study aimed to determine the optimal postsurgical surveillance strategy for stage II/III GC patients and compare its cost-effectiveness with traditional surveillance strategies.

DETAILED DESCRIPTION:
Background The development of existing follow-up strategies is mainly based on experts' consensus and researches on recurrence patterns due to the lack of direct evidence and unified standards. On the one hand, it is unreasonable to carry out the same postsurgical surveillance for all stage II/III GC patients. Additionally, In addition to the early detection of recurrence, the optimal follow-up strategy should also balance cost and effectiveness. There were no criteria for the arrangement of follow-up in different guidelines, and the optimal postoperative follow-up strategy for patients with stage II/III GC remains unclear.

Methods Prospectively collected data from stage II/III GC patients (n=1,661) who underwent gastrectomy at Fujian Medical University Union Hospital (FJMUUH) between January 2010 and October 2015. For external validation, two independent cohorts were included, which were composed of 380 stage II/III GC patients who underwent gastrectomy at the Mayo Clinic between July 1991 and July 2012 and 270 stage II/III GC patients at the Qinghai university affiliated hospital (QUAH) between May 2010 and Oct 2014. Random survival forest models were used to predict dynamic recurrence hazards and to construct individual surveillance strategies for stage II/III GC. Cost-effectiveness were assessed by Markov model.

ELIGIBILITY:
Inclusion Criteria:

* (1) Eastern Cooperative Oncology Group (ECOG) scores of 0 (asymptomatic) or 1 (symptomatic but completely ambulatory); (2) pathologically confirmed AGC (pStage II and III, except pT4b); (3) no distant metastasis or invasion of adjacent organs (e.g., pancreas, spleen, liver, and colon) detected intra- or post-operatively; and (4) D2 lymph node dissection of gastric cancer.

Exclusion Criteria:

* (1) American Society of Anesthesiologists (ASA) grade >2; (2) remnant gastric or neuroendocrine cancer; (3) history of neoadjuvant chemotherapy; (4) palliative surgery; and (5) death within 30 days after surgery.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A total of 1,661 stage II/III GC patients who underwent gastrectomy at Fujian Medical University Union Hospital (FJMUUH) between January 2010 and October 2015. For external validation, two independent cohorts were included, which were composed of 380 stage II/III GC patients who underwent gastrectomy at the Mayo Clinic between July 1991 and July 2012 and 270 stage II/III GC patients at the Qinghai university affiliated hospital (QUAH) between May 2010 and Oct 2014.
Sampling Method: Non-Probability Sample
Enrollment: 2311 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
recurrence rate | 5 years
  distant, peritoneal, and local recurrence

SECONDARY OUTCOMES:
Delayed-detection months | 5 years
  A hypothetical cohort of 1000 GC patients was generated to compare the effectiveness of surveillance among the above-mentioned strategies by calculating the sum of the delayed detection months. Delayed detection months were defined as the duration from the occurrence of failure to the next-nearest follow-up. For instance, if a patient develops distant metastasis in the 3rd month while the next nearest planned visit is in the 5th month, the delayed -detection time for this patient is 2 months. The total number of delayed detection months of our risk-based surveillance schedule and that of the control strategies were simulated and compared.
Incremental cost-effectiveness ratios (ICERs) | 5 years
  incremental cost-effectiveness ratios (ICERs) were calculated by dividing the difference in cost by the difference in QALY.

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, MD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Department of Gastric Surgery, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wu D, Lu J, Lin J, Xu BB, Xue Z, Zheng HL, Lin GS, Huang JB, Shen LL, Zheng CH, Li P, Xie JW, Wang JB, Lin JX, Chen QY, Cao LL, Ma YB, Truty MJ, Huang CM. An international multi-institution real-world study of the optimal surveillance frequency for stage II/III gastric cancer: the more, the better? Int J Surg. 2023 Dec 1;109(12):4101-4112. doi: 10.1097/JS9.0000000000000731. PMID 37800589